CLINICAL TRIAL: NCT01755650
Title: A Phase 0 Exploratory Microdosing Study of S-(3-18Ffluoropropyl)Homocysteine Hydrochloride; 18FFPM Using PET/CT in Patients With a Variety of Malignancies.
Brief Title: Phase 0 of 18F FPM Using PET/CT in Patients With a Variety of Malignancies
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: 6 patients were recuited. Due to inability of the tracer to detect regions of interest sufficiently, the trial was closed early.
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 11/31
Record Dates: First submitted 2012-12-16; First posted 2012-12-24 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Squamous Cell Carcinoma
Keywords: 18F FPM; PET/CT; microdosing
MeSH Terms: conditions — Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D-18F FPM (Experimental)
  Interventions: Radiation: 18F FPM
- L-18F FPM (Experimental)
  Interventions: Radiation: 18F FPM

INTERVENTIONS:
Radiation: 18F FPM

SUMMARY:
The purpose of this study is to investigate the safety and potential effectiveness of the imaging compound 18F FPM for finding sites of malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to any protocol-specific procedures
* Male and female patients with histologically confirmed squamous cell carcinoma
* At least one site of active malignancy, as demonstrated on the pre-study 18F FDG PET/CT scan performed as part of routine clinical care
* Age >/= 18 years
* Life expectancy >/= 3 months
* ECOG Performance score of 0-2

Exclusion Criteria:

* Pregnant or breastfeeding females
* Systemic anti-neoplastic therapy within the 2 weeks prior to the pre-study 18F FDG PET/CT scan until after the 18F FPM PET/CT scan
* Any serious medical condition which the investigator feels may interfere with the procedures or evaluations of the study
* Patients unwilling or unable to comply with protocol or with a history of non-compliance or inability to grant informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2017-11-03 (Actual); Study Completion 2017-11-03 (Actual)

PRIMARY OUTCOMES:
Safety of D-18F FPM and L-18F FPM administration as measured by occurrence of adverse clinical, biochemical or haematological events following 18F FPM administration | Up to 28 days following 18F FPM administration (+/- 7 days)

SECONDARY OUTCOMES:
Percentage of injected D-18F FPM and L-18F FPM dose in organs of interest. | 10, 30, 60 and 120 minutes post 18F FPM administration
Percentage of unmetabolized D-18F FPM and L-18F FPM in plasma and urine after radiotracer administration. | 30 (plasma only) and 90 (plasma and urine) minutes post 18F FPM administration
Absorbed organ doses expressed as micro Sv/MBq of administered D-18F FPM and L-18F FPM, and whole body dose expressed as milliSv/200MBq of administered dose | 10, 30, 60 and 120 minutes post 18F FPM administration

CONTACTS AND LOCATIONS:
Overall Officials: Ben Solomon, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Centre, East Melbourne, Victoria, Australia